CLINICAL TRIAL: NCT02305303
Title: Impact of an Intensive Care Unit Diary on Long-term Quality of Life After Severe Trauma
Brief Title: Diary for Severe Trauma
Acronym: Qualitrau
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K131202
Record Dates: First submitted 2014-09-09; First posted 2014-12-02 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Quality of life; post-traumatic stress disorder; trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diary (Experimental): Use of diary
  Interventions: Procedure: Diary
- Without Diary (No Intervention)

INTERVENTIONS:
Procedure: Diary — A diary written prospectively during the ICU stay by the staff and relatives
  Arms: Diary

SUMMARY:
Treatment of severe trauma patients includes intensive cares. Both trauma and intensive care may lead to a post-traumatic stress disorder‬ and then to a decreased quality of life. Diaries may improve the frequency and the intensity of PTSD. Aim of investigator is to assess if diaries may improve quality of life after a severe trauma.

DETAILED DESCRIPTION:
Trauma is the third cause of death in France and the first cause of death of people under 40 years (48 000 deaths a year).

Severe trauma defined by an Injury Severity Score ( ISS) > 15 implies intensive care.

Intensive care unit admission induces considerable psychological distress and memory troubles, both promoting posttraumatic stress disorder (PTSD) and symptoms of anxiety and depression. A diary written prospectively during the ICU stay by the staff and relatives has been suggested as a means of help¬ing patients to build a more detailed and factual narrative of their ICU stay than would be possible based only on their fragmented memories. Garrouste et al. have shown that the intensive care unit diary significantly affected posttraumatic stress disorders in surviving patients 12 months after intensive care unit discharge.

Besides, severe trauma by itself may decrease the quality of life (QoL). It is recommended to assess QoL on one year after the trauma. In trauma patients, the change in QoL is associated with the presence of a PTSD.

Consequently, severe trauma patients who undergo a double stress, that of the accident and that of the intensive care unit stay: they may so even more have a decrease of their QoL by developing a PSTD.

The investigator formulate the hypothesis that a diary, written by the staff and relatives from the very acute phase of the ICU stay (first 48 hours) to the discharge of ICU would improve the QoL and would decrease the frequency and the intensity of PTSD of the severe trauma patients one year after the trauma.

ELIGIBILITY:
Inclusion Criteria:

* all patients over 18
* with severe trauma (Injury Severity Score (ISS) > 15)
* admitted in our trauma centered and hospitalized in intensive care unit for more than 48 h

Exclusion Criteria:

* non-French language fluent patients
* Patients with dementia
* Hospitalization in intensive care unit less than
* opposition to data utilization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2014-11-09 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Quality of life | 12 months after the trauma
  To assess the quality of life (QoL), investigator will use the WHO Quality of Life questionnaire Brief Version (WHOQOL- Bref) in its french-language version. exploring four dimensions (physical, psychological, social and environmental).

SECONDARY OUTCOMES:
post-traumatic stress disorder (PTSD) | 12 months after the trauma
  To assess the frequency and the intensity of PTSD, investigator will use the Impact of Events Scale-revised questionnaire (IES-R), a valid and reliable 22-item screening tool that assesses symptoms of intrusion, avoid-ance, and hyperarousal
predictive factors of decrease in QoL after severe trauma | 12 months after the trauma
  At the admission, investigator will notice trauma data. Plus, the investigator will ask the conscious patient or his/her next of kin about sociodemographic, professional characteristics at the admission and 12 months after the trauma
patients' expectations | 12 months after the trauma
  Conduction of a quality study through a semi-open questionary about the care during and after the intensive care unit stay and about the diary (experimental group only)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Benazzour, Nurse, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Département d'Anesthésie-Réanimation Groupe Hospitalier Pitié Salpêtrière, Paris, France